CLINICAL TRIAL: NCT00589667
Title: A Phase II Study of Pemetrexed Plus Gemcitabine for Metastatic/Recurrent Head and Neck Cancer (HNSCC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-087
Record Dates: First submitted 2007-12-26; First posted 2008-01-10 (Estimated); Results first posted 2014-03-05 (Estimated); Last update posted 2014-04-02 (Estimated); Status verified 2014-03

CONDITIONS: Head and Neck Cancer
Keywords: Head and Neck Cancer; GEMCITABINE; PEMETREXED; ALTIMA; epidermoid/squamous cell; carcinoma; pharynx; larynx; paranasal sinus; head/neck squamous cell carcinoma
MeSH Terms: conditions — Head and Neck Neoplasms; Carcinoma; Laryngeal Diseases; Squamous Cell Carcinoma of Head and Neck | interventions — Pemetrexed; Gemcitabine

ARMS (1):
- Treatment (Experimental): Patients will receive pemetrexed (500 mg/m2 IV infusion over approximately 10 minutes) followed immediately by gemcitabine (1250 mg/m2 IV infusion given over approximately 30 minutes) on day 1 and day 15 of a 28-day cycle.
  Interventions: Drug: Pemetrexed plus Gemcitabine

INTERVENTIONS:
Drug: Pemetrexed plus Gemcitabine — Patients will receive pemetrexed (500 mg/m2 IV infusion over approximately 10 minutes) followed immediately by gemcitabine (1250 mg/m2 IV infusion given over approximately 30 minutes) on day 1 and day 15 of a 28-day cycle. Vitamin supplementation will be as follows: Vitamin B12: 1000 µg IM injection no less than 1 week prior to the first dose of pemetrexed, and continuing approximately every 9 weeks until 3 weeks after the last dose of pemetrexed.
  Folic acid: The preferred oral daily dose of folic acid is 350 to 1000 µg. Daily folate supplementation begins no less than 1 week prior to the first dose of pemetrexed and continues until 3 weeks after the last dose of pemetrexed.
  For rash prophylaxis, dexamethasone (4 mg po twice per day) should be taken on the day before, the day of, and the day after each dose of pemetrexed unless clinical contraindications exist.
  Other Names: Alimta; LY231514

SUMMARY:
The purpose of this study is to determine if the combination of 2 chemotherapy drugs called pemetrexed and gemcitabine might be effective treatment for head and neck squamous cell cancer. The researchers want to find out what effects, good and/or bad, that this treatment has on head and neck cancer.

DETAILED DESCRIPTION:
Pemetrexed (500 mg/m2) and gemcitabine (1250 mg/m2) will be given together on Days 1 and 15 of a 28 day cycle in patients with recurrent or metastatic head and neck squamous cell carcinoma (HNSCC). Patients will not have received more than 2 prior chemotherapy regimens in the recurrent/metastatic disease setting. Vitamin B12 and folate supplementation will be administered per standard guidelines for pemetrexed chemotherapy.

The primary endpoint is the objective radiologic response rate. Radiologic imaging of evaluable disease will take place after every 2 cycles. Patients may remain on study until progression of disease or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have microscopically confirmed epidermoid/squamous cell carcinoma (HNSCC) of the oral cavity, pharynx, larynx, paranasal sinus, or head/neck squamous cell carcinoma unknown primary.
* Patients must have recurrent or metastatic disease which is not amenable to curative-intent therapy with surgery or radiation.
* No more than 2 prior cytotoxic therapies in the recurrent or metastatic disease setting are permitted.
* Patients must be at least 18 years of age.
* Karnofsky Performance status must be ≥ 70%.
* Disease must be measurable by RECIST criteria.
* At least 4 weeks must have elapsed from previous radiation therapy. Patient must have recovered from the acute toxic effects of treatment prior to study enrollment.
* Prior radiation therapy to ≤ 25% of bone marrow is allowed. Prior radiation to the whole pelvis and/or brain is not allowed.
* Adequate organ function
* Patients of childbearing potential must have a negative test for pregnancy at time of enrollment based on a urine or serum pregnancy test. Patients must agree to use a reliable method of birth control during and for 3 months following the last dose of study drug.
* Patient must reside in geographic proximity to MSKCC for adequate follow-up during treatment, per investigator discretion.
* Patients must sign an informed consent document.

Exclusion Criteria:

* Previous exposure to pemetrexed (Alimta) or gemcitabine (Gemzar).
* Pregnancy or breast-feeding.
* Serious concomitant systemic disorders (for example, active infection) that, in the opinion of the investigator, would compromise the safety of the patient or compromise the patient's ability to complete the study.
* History of any brain metastases.
* Inability or unwillingness to take folic acid, vitamin B12 supplementation, or dexamethasone.
* Patients will be excluded if they will be unable to hold use of nonsteroidal antiinflammatory agents (NSAIDS) with short elimination half lives

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2006-09; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David G Pfister, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering web site — http://www.mskcc.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Protocol Open to Accrual 09/08/1998 Protocol Closed to Accrual 07/22/2008 Primary Completion Date 07/13/2010 Recruitment Location is the medical clinic.
Groups:
- Pemetrexed Plus Gemcitabine: Patients will receive pemetrexed (500 mg/m2 IV infusion over approximately 10 minutes) followed immediately by gemcitabine (1250 mg/m2 IV infusion given over approximately 30 minutes) on day 1 and day 15 of a 28-day cycle.
Period: Overall Study
Arm/Group | Pemetrexed Plus Gemcitabine
Started | 26
Completed | 23
Not Completed | 3
Not completed — Adverse Event | 2
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Pemetrexed Plus Gemcitabine
Number analyzed (Participants) | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.5 (43.13351365)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 20
Region of Enrollment [Number; unit: participants]
  United States | 26

OUTCOME MEASURES:

1. Primary Outcome: Overall Objective Response
Description: To determine the objective radiologic response rate of pemetrexed and gemcitabine in patients with recurrent or metastatic Head and Neck Squamouse Cell Carcinoma.
  Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 2 years
Population: All assessable patients as indicated in the protocol.
Measure: Number; unit: participants
Arm/Group | Pemetrexed Plus Gemcitabine
Number analyzed (Participants) | 25
participants
  Partial Response | 4
  Stable Disease | 18
  Progression of Disease | 2
  Response not available | 1

2. Secondary Outcome: Median Overall Survival
Description: To determine the median overall survival for patients with recurrent or metastatic Head and Neck Squamous Cell Carcinoma treated with pemetrexed and gemcitabine.
Time Frame: 2 years
Population: There were 25 assessable patients as described in the protocol.
Measure: Median (Full Range); unit: months
Arm/Group | Pemetrexed Plus Gemcitabine
Number analyzed (Participants) | 25
months | 8.8 [1.9 to 30.9]

ADVERSE EVENTS:
Arm/Group | Pemetrexed Plus Gemcitabine
Serious Adverse Events (participants affected / at risk) | 12/25
Other Adverse Events (participants affected / at risk) | 23/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pemetrexed Plus Gemcitabine (N=25)
Hyponatremia (Metabolism and nutrition disorders) | 3 (4)
Immune system disorder (Immune system disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 3 (5)
Confusion (Psychiatric disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (5)
Edema-Head and Neck (General disorders) | 1 (2)
Edema-limb (General disorders) | 1 (1)
Fatigue (General disorders) | 2 (3)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Fever (General disorders) | 2 (3)
Hemoglobin (Investigations) | 2 (2)
Hypotension (Vascular disorders) | 2 (3)
Skin Infection (Infections and infestations) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
Mucositis-esophagus (Gastrointestinal disorders) | 1 (1)
Neutrophil count decrease (Investigations) | 3 (3)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (2)
Psychosis (Psychiatric disorders) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Thrombosis (Vascular disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pemetrexed Plus Gemcitabine (N=25)
Alanine aminotransferase increased (Investigations) | 2 (2)
Fatigue (General disorders) | 3 (3)
Anemia (Blood and lymphatic system disorders) | 10 (51)
INR increased (Investigations) | 2 (19)
White blood cell decreased (Investigations) | 5 (26)
Lymphocyte count decreased (Investigations) | 20 (166)
Neutrophil count decreased (Investigations) | 3 (13)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (7)
Platelet count decreased (Investigations) | 2 (11)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes